CLINICAL TRIAL: NCT07114211
Title: A Real-world Observational Study on the Diagnostic Value of 99mTc-FAPI Quantitative SPECT/CT Imaging in Adult Solitary Bone Lesions
Brief Title: A Study on the Diagnostic Value of 99mTc-FAPI Quantitative SPECT/CT Imaging in Adult Solitary Bone Lesions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KY20252270
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Bone Lesion; SPECT-CT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 99mTc-HYNIC-FAPI-04 group (Experimental)
  Interventions: Diagnostic Test: 99mTc-HYNIC-FAPI-04 SPECT-CT

INTERVENTIONS:
Diagnostic Test: 99mTc-HYNIC-FAPI-04 SPECT-CT — Perform quantitative SPECT/CT with 99mTc-HYNIC-FAPI-04 on selected patients. Acquire whole-body images in a planar format and SPECT/CT images of two or more sites in a tomographic format.

SUMMARY:
Using the novel FAPI probe 99mTc-HYNIC-FAPI-04 and quantitative SPECT/CT imaging technology, this study investigates the diagnostic efficacy of 99mTc-HYNIC-FAPI-04 quantitative SPECT/CT in patients with common solitary bone lesions in adults, and compares its diagnostic performance with conventional CT, MRI, and 99mTc-MDP bone scintigraphy. Follow-up pathological results of patients post-surgery were analysed to assess the accuracy of 99mTc-HYNIC-FAPI-04 diagnostic outcomes, and its diagnostic value and significance were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Benign solitary bone lesions in adults (fibrous cortical defects, fibrous hyperplasia, non-ossifying fibroma, osteoblastoma, osteoid osteoma, osteochondroma, etc.); Malignant solitary bone lesions in adults (osteosarcoma, Ewing's sarcoma, chondrosarcoma, malignant giant cell tumour of bone, etc.); Other fibroblast-rich bone lesions (chordoma, alveolar soft part sarcoma, fibrosarcoma, malignant fibrous histiocytoma, etc.).

Exclusion Criteria:

* Severe liver and kidney dysfunction; Pregnant women and breastfeeding patients; Patients in poor physical condition who cannot tolerate the examination; Patients who cannot cooperate to complete the examination; Patients under the age of 18.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
SUVmax | 1 day from injection of the tracer
  Maximum standardised intake value
SUVmean | 1 day from injection of the tracer
  Average standardised intake value

IPD SHARING:
Plan to Share IPD: No